CLINICAL TRIAL: NCT05869591
Title: Pharmacokinetics and Pharmacodynamics Assessment of Apixaban and Edoxaban in Patients with Child a or B Liver Cirrhosis
Brief Title: DOAC in Patients with Child a or B Liver Cirrhosis
Acronym: CIRROAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Lorenzo ALBERIO, Prof Dr. méd, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CER-VD 2022-01395
Record Dates: First submitted 2023-05-03; First posted 2023-05-22 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Liver Cirrhosis
Keywords: Cirrhosis; DOAC; Thrombin generation; Anticoagulation
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — apixaban; edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cirrhotic patients with Child A or B under apixaban (Experimental): Twenty non-anticoagulated patients with Child A or B liver cirrhosis will receive a therapeutic dose of apixaban (Eliquis®) for 7 consecutive days.
  Blood samples will be collected just before and after apixban intake at day 1 and 3. Another blood samples are collected at day 8 and at day 9.
  In vivo thrombin generation parameters (F1+2, TAT, fibrin monomers, D-dimers), ex vivo thrombin generation parameters [ST Genesia (Drugscreen)], as well as peak and trough apixaban levels will be measured.
  Interventions: Drug: Apixaban 5 MG [Eliquis]
- Cirrrhotic patients with Child A or B under edoxaban (Experimental): Twenty non-anticoagulated patients with Child A or B liver cirrhosis will receive a therapeutic dose of edoxaban (Lixiana®) for 7 consecutive days.
  Blood samples will be collected just before and after edoxaban intake at day 1 and 3. Another blood samples are collected at day 8 and at day 9.
  In vivo thrombin generation parameters (F1+2, TAT, fibrin monomers, D-dimers), ex vivo thrombin generation parameters [ST Genesia (Drugscreen)], as well as peak and trough edoxaban levels will be measured.
  Interventions: Drug: Edoxaban 60 MG [Lixiana]

INTERVENTIONS:
Drug: Apixaban 5 MG [Eliquis] — Pharmacokinetics and pharmacodynamics assessment of apixaban in patients with Child A or B liver cirrhosis
  Arms: Cirrhotic patients with Child A or B under apixaban
Drug: Edoxaban 60 MG [Lixiana] — Pharmacokinetics and pharmacodynamics assessment of edoxaban in patients with Child A or B liver cirrhosis
  Arms: Cirrrhotic patients with Child A or B under edoxaban

SUMMARY:
The goal of this clinical trial is to investigate pharmacokinetics and pharmacodynamics of direct oral anticoagulant drugs (DOAC), specifically apixaban and edoxaban, in patients with Child A or B liver cirrhosis (LC). The primary objective of this study is to verify the ability of apixaban and edoxaban to decrease in vivo thrombin generation in LC patients.

Participants will be randomly assigned to either apixaban (Eliquis®) or edoxaban (Lixiana®) at a therapeutic dosage for 7 consecutive days.

The results of this investigation will contribute to designing a prospective multicentre interventional study to investigate the efficacy of DOAC to improve clinical outcomes in patients with LC

DETAILED DESCRIPTION:
Patients with liver cirrhosis (LC) have a higher risk to develop venous thromboembolism (VTE), in particular portal vein thrombosis (PVT) and the risk is increased with advanced liver disease. Some studies have shown that anticoagulant therapy in patients with LC and PVT could improve their prognosis by reducing liver decompensation, variceal bleeding, encephalopathy, and portal hypertension complications. Direct oral anticoagulant drugs (DOAC) seem to be as effective and safe as traditional anticoagulant drugs [vitamin K antagonists (VKA) and low molecular weight heparins (LMWH)]. Moreover, some studies showed lower bleeding rate and more recanalization of PVT with DOAC than traditional anticoagulant drugs. However, physicians are still reluctant to anticoagulate this population. This is well illustrated by the lower rate of adequate prophylaxis during in-hospital treatment in LC compared to other patients. This is probably due to two reasons. First, the fear of inducing bleeding in patients with increased INR and persistent thrombocytopenia, although it has been shown that the VTE risk is independent of INR and thrombocytopenia. Second, there is still a large knowledge gap on the effects of the various anticoagulant drugs and on the best anticoagulant molecule to employ in this population. Indeed, both VKA and LMWH present several disadvantages in LC patients. VKA are not recommended because of unreliable INR (already increased at baseline) and the risk of pseudo-therapeutic INR values. As for LMWH, a non-negligible increase of bleeding complications has been observed in LC patients. It has been demonstrated that patients with LC exhibit a lower anti-Xa activity when treated with LMWH compared to other patients and that after spiking their plasma with a given amount of LMWH, the measured anti-Xa activity was lower than in plasma from healthy controls. Of note, the anti-Xa activity was corrected after supplementation of antithrombin. In case of anti-Xa monitoring, this could lead to LMWH overdosing. In fact, despite a lower anti-Xa activity, the anticoagulant effect of LMWH seems to be increased in LC patients when assessed by thrombin generation, possibly because of antithrombin-independent antithrombotic actions of LMWH. Therefore, also LMWH are not ideal for LC patients. Nevertheless, both VKA and LMWH are the anticoagulant most frequently administrated to patients with LC, possibly also because of limited data about DOAC. In fact, patients with advanced liver disease or "hepatic coagulopathies" have been excluded from clinical trials investigating DOAC.

DOAC (apixaban, rivaroxaban, edoxaban, and dabigatran) represent an alternative to VKA and LMWH with specific advantages, particularly the oral intake and a direct action on coagulation factors. Different studies showed similar to lower bleeding rates in cirrhotic patients on DOAC compared to cirrhotic patients treated with warfarin or heparins. This suggests that DOAC are possibly a safe and effective alternative to VKA and LMWH. However, before performing large randomised controlled trials, the effect of specific DOAC in LC should be further studied, to select the ideal molecule.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient with previously diagnosed liver cirrhosis Child A or B
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Oesophageal varices with grade superior to 1 or with red signs
* Active ulcer disease of the gastrointestinal tract
* History of haemorrhagic stroke
* Severe uncontrolled hypertension
* Recent brain, spinal or ophthalmic surgery
* Kidney function inadequate for DOAC treatment
* Concomitant treatment with anti-platelet drugs
* Concomitant treatment with anticoagulant drugs (VKA, LMWH, DOAC)
* Any contraindications for DOAC administration
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes from thrombin generation parameters before and after apixaban (Eliquis®) intake | At day 1 and day 3 before DOAC intake and 2 hours after intake. At day 8, 24 hours after last pill intake.
  Global thrombin generation assay will be performed using ST Genesia (Stago, Asnière-sur-Seine, France) with Drugscreen reagents (high tissue factor concentration) will be used and all thrombin generation parameters will be retrieved.
Changes from thrombin generation parameters before and after edoxaban (Lixiana®) intake | At day 1 and day 3 before DOAC intake and 2 hours after intake. At day 8, 24 hours after last pill intake.
  Global thrombin generation assay will be performed using ST Genesia (Stago, Asnière-sur-Seine, France) with Drugscreen reagents (high tissue factor concentration) will be used and all thrombin generation parameters will be retrieved.
Changes from peak and trough levels of apixaban (Eliquis ®) | At day 1, at peak level (2 hours after intake). At day 3, at steady state (before intake) and at peak level (2 hours after intake). A day 8 at residual concentration (24 hours after last pill intake). At day 9, 48 hours after last intake.
  Concentration of DOAC will be assessed with specific anti-Xa assays using Sysmex CS5100 coagulation analyser (Siemens Healthcare, Erlangen, Germany) and reagents: Hyphen Biophen® Heparin (Hyphen BioMed, Neuville-sur-Oise, France).
Changes from peak and trough levels of edoxaban (Lixiana ®) | At day 1, at peak level (2 hours after intake). At day 3, at steady state (before intake) and at peak level (2 hours after intake). A day 8 at residual concentration (24 hours after last pill intake). At day 9, 48 hours after last intake.
  Concentration of DOAC will be assessed with specific anti-Xa assays using Sysmex CS5100 coagulation analyser (Siemens Healthcare, Erlangen, Germany) and reagents: Hyphen Biophen® Heparin (Hyphen BioMed, Neuville-sur-Oise, France).

SECONDARY OUTCOMES:
Changes from Thrombin-antithrombin complex (TAT) concentration before and after intake of apixaban (Eliquis®) for one week in patients with Child A or B liver cirrhosis. | At day 1 and day 3 before DOAC intake and 2 hours after intake. At day 8, 24 hours after last DOAC pill intake.
  In vivo markers of coagulation as TAT (in ng/ml) will be measured by a quantitative enzyme immunoassay (ELISA), according to the protocol of the manufactures (Enzygnost® TAT micro Siemens). The absorbance will be measured using a Dynex microplate reader at 450 nm.
Changes from Thrombin-antithrombin complex (TAT) concentration before and after intake of edoxaban (Lixiana ®) for one week in patients with Child A or B liver cirrhosis. | At day 1 and day 3 before DOAC intake and 2 hours after intake. At day 8, 24 hours after last DOAC pill intake.
  In vivo markers of coagulation as TAT (in ng/ml) will be measured by a quantitative enzyme immunoassay (ELISA), according to the protocol of the manufactures (Enzygnost® TAT micro Siemens). The absorbance will be measured using a Dynex microplate reader at 450 nm.
Changes from prothrombin activation fragments 1+2 (F1+2) concentration before and after intake of apixaban (Eliquis®) for one week in patients with Child A or B liver cirrhosis. | At day 1 and day 3 before DOAC intake and 2 hours after intake. At day 8, 24 hours after last DOAC pill intake.
  In vivo markers of coagulation as F1+2 (in pmol/l) will be measured by a quantitative enzyme immunoassay (ELISA), according to the protocol of the manufactures (Enzygnost® F1+2 micro Siemens). The absorbance will be measured using a Dynex microplate reader at 492 nm.
Changes from prothrombin activation fragments 1+2 (F1+2) concentration before and after intake of edoxaban (Lixiana®) for one week in patients with Child A or B liver cirrhosis. | At day 1 and day 3 before DOAC intake and 2 hours after intake. At day 8, 24 hours after last DOAC pill intake.
  In vivo markers of coagulation as F1+2 (in pmol/l) will be measured by a quantitative enzyme immunoassay (ELISA), according to the protocol of the manufactures (Enzygnost® F1+2 micro Siemens). The absorbance will be measured using a Dynex microplate reader at 492 nm.
Changes from D-dimers concentration before and after intake of apixaban (Eliquis®) for one week in patients with Child A or B liver cirrhosis. | At day 1 and day 3 before DOAC intake and 2 hours after intake. At day 8, 24 hours after last DOAC pill intake.
  D-Dimers concentrations (in ng/ml) will be measured by an automated quantitative immunoassay, according to the manufacturer's instructions (INNOVANCE® D-dimer).
Changes from D-dimers concentration before and after intake of edoxaban (Lixiana®) for one week in patients with Child A or B liver cirrhosis. | At day 1 and day 3 before DOAC intake and 2 hours after intake. At day 8, 24 hours after last DOAC pill intake.
  D-Dimers concentrations (in ng/ml) will be measured by an automated quantitative immunoassay, according to the manufacturer's instructions (INNOVANCE® D-dimer).
Safety analysis with the identification of specific AEs and SAEs | From day 1 to day 14.
  Major and clinically relevant bleeding events will be retrieved.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Alberio, Prof Dr. med, Principal Investigator — CHUV
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No